CLINICAL TRIAL: NCT05033015
Title: Effect of an Enzyme-containing Mouth Rinse on Dental Biofilm Accumulation in Patients With Fixed Orthodontic Appliances: a Randomized Placebo-controlled Clinical Trial
Brief Title: Effect of Enzyme-containing Mouth Rinse on Dental Biofilm in Patients With Fixed Orthodontic Appliances
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Malmö University (Other)
Collaborators: Novozymes A/S (Industry)
Responsible Party: Principal Investigator, Mikael Sonesson, Associate Professor, Malmö University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2020-05221
Record Dates: First submitted 2021-08-27; First posted 2021-09-02 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Caries
MeSH Terms: interventions — Mouthwashes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Self applied
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test (Experimental): Mouth rinse containing enzymes
  Interventions: Procedure: Mouth rinse
- Placebo (Active Comparator): Control, same content as test, without enzymes
  Interventions: Procedure: Mouth rinse

INTERVENTIONS:
Procedure: Mouth rinse — To test a novel mouth rinse containing enzymes to prevent development of WSL with a control

SUMMARY:
Caries is a biofilm-mediated global public health problem causing health, social and economic consequences for individuals, communities and countries.

Treatment with fixed orthodontic appliances is associated with impaired oral hygiene. This results in a demineralization of the enamel (white spot lesions). The prevalence is fairly high (30-50%) among adolescents and self-applied fluorides cannot completely prevent such lesions. It is therefore important to investigate novel approaches to combat these unwanted adverse effects. A systematic review has suggested that mouthwashes may be suitable technology to control biofilm accumulation in orthodontic patients. The aim of the present pilot study is to evaluate the effect of a novel mouth rinse containing a blend of natural enzymes in addition to fluoride on the presence of oral biofilm in patients undergoing treatment with fixed orthodontic appliances.

DETAILED DESCRIPTION:
Study design A randomized, double-blind placebo-controlled design with two parallel groups will be performed. The null hypothesis is that the effect on the dental biofilm of the experimental mouth rinse will not differ from that of a placebo rinse without active enzymes.

Patients Adolescent patients (14-18 years) attending the Orthodontic specialist clinic in Karlshamn, Sweden will be invited.

Methods The patients are randomly allocated to the test group or the control group with aid of computer-generated random number. After the baseline clinical registration, the participants are instructed to thoroughly rinse their mouth by swishing the mouth rinse around the teeth twice daily (morning and evening) for 30 seconds. 10 mL of the assigned solution should be used at each occasion. After rinsing, the subjects should spit out but no additional rinsing with water is allowed afterwards. The duration of the intervention is one week and the patients are instructed to brush their teeth twice daily using a 1,450 ppm fluoride toothpaste. The test and the placebo mouth rinses should be separated from the daily tooth brushing with at least 30 minutes. The patients are provided with a standardized enzyme-free toothpaste to be used during the intervention.

Intervention The water-based test rinse contains a blend of enzymes in an aqueous solution. The safety evaluation of the three enzymes is tested. The control (placebo) rinse has an identical taste, color and texture but contains no enzymes. The solutions are provided in color-coded tubes, each containing exactly 10 mL of the test or placebo mouth rinse. An independent monitor based at Malmö University but not involved in the project will guarantee the allocation concealment.

Statistical methods All clinical data are processed with the IBM-SPSS software (version 25.0, Chicago, USA). Descriptive analyses will be performed with continuous and categorical data. Differences between and within the groups are compared with unpaired and paired tests, respectively. A p-value less than 0.05 is regarded as statistically significant. The statistical calculations are completed before the group allocation is unveiled.

Power calculation There are no previous clinical data available on the biofilm response to the experimental mouth rinse and this pilot study will form the basis of future sample-size calculations. A mean difference of 0.5 units (SD 0.4) is considered as clinically meaningful and an estimation based on α=0.05 and β=0.8 indicate that 20 patients in each group needs to be enrolled to the pilot project.

ELIGIBILITY:
Inclusion Criteria:

* patients with fixed orthodontic appliances in at least one arch for at least 3-6 months,
* visible plaque around the bracket bases of at least 6 teeth
* repeated oral hygiene instructions have been given during the orthodontic treatment

Exclusion Criteria:

* clinically visible active caries lesions and/or periodontitis
* significant oral soft tissue pathology based on a visual examination
* history of allergy or significant adverse events following use of oral hygiene products such as toothpastes, mouth rinses, breath mints, lozenges, or chewing gum or their ingredients
* history of allergies to ingredients in the test product, including allergy against enzymes
* history of common food allergies, such as peanuts, tree nuts, milk, eggs, shellfish, fish, wheat, soybeans
* self-reported serious medical conditions, pregnancy or nursing
* acute sinusitis or severe oral-pharyngeal infections

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-12-07 (Estimated)

PRIMARY OUTCOMES:
dental biofilm in test and control | 7 days
  clinical scoring according to Orthodontic Plaque Index, of the amount and extension of the dental biofilm at baseline and after 7 days. Score 0 no extension Score 5 extended biofilm

SECONDARY OUTCOMES:
composition of the salivary microbiome | 7 days
  DNA-extraction and whole genome sequencing will be conducted when all samples are collected. The DNA-extraction will be performed with Macherey-Nagel™ NucleoSpin™ Soil kit. The V3-V4 region of 16S will be PCR amplified using universal primers and sequenced using Illumina MiSeq 300bp paired end.
  DNA-extraction and whole genome sequencing will be conducted when all samples are collected. The DNA-extraction will be performed with Macherey-Nagel™ NucleoSpin™ Soil kit. The V3-V4 region of 16S will be PCR amplified using universal primers and sequenced using Illumina MiSeq 300bp paired end.

CONTACTS AND LOCATIONS:
Overall Officials: Mikael Sonesson, Assoc Prof., Principal Investigator — Malmö University
Locations (1):
- Mikael Sonesson, Malmo, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hoffstedt T, Skov Hansen LB, Twetman S, Sonesson M. Effect of an enzyme-containing mouthwash on the dental biofilm and salivary microbiome in patients with fixed orthodontic appliances: a randomized placebo-controlled pilot trial. Eur J Orthod. 2023 Feb 10;45(1):96-102. doi: 10.1093/ejo/cjac062. PMID 36214729